CLINICAL TRIAL: NCT06801782
Title: Effectiveness of Attention/executivefunctions Training on Prospective Memory Abilities of Parkinson's Disease Subjects with Mild Cognitive Impairment and Healthy Aged Individuals: a Placebo-controlled Study with a Combined Immersive Virtual Reality and Telemedicine Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Silvia Zabberoni, Researcher Psychologist, PhD, Princial Investigator, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE/PROG.758
Record Dates: First submitted 2025-01-17; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Parkinson's Disease with Cognitive Impairment; Healthy Elderly
Keywords: placebo controlled trial; Cognitive training; Prospective Memory; Virtual reality; Telemedicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive executive functions training implemented in immersive virtual reality, remotly delivered (Experimental): The training group (TR-C) underwent a 4-week immersive virtual reality (iVR) program designed to improve planning, shifting, and updating skills to enhance prospective memory (PM) in PD-MCI patients. Participants completed 12 sessions of 30 minutes each in a virtual supermarket, performing tasks that strengthened executive functions. The planning task involved planning a route to purchase items, the shifting task required alternating between product categories, and the updating task was based on a memory recall of objects. Each task had 10 levels, progressively increasing in difficulty, with participants advancing after completing three consecutive successful trials, receiving feedback at each level.
  Interventions: Behavioral: Experimental Cognitive training in Immersive Virtual Reality and Telemedicine approach
- Active Placebo implemented in immersive virtual reality, remotly delivered (Active Comparator): The active placebo group shared the same virtual environment and interaction methods as the training group (Arm 1), using the Oculus Go and remote telemedicine. This condition involved tasks with low cognitive demands, similar to everyday activities. The placebo-planning task required following a fixed shopping list order, the placebo-shifting task involved quickly selecting items from the shelves, and the placebo-updating task required remembering the last item from a conveyor belt sequence. The frequency, duration, and number of levels and trials were identical to the training condition (3 sessions per week, 30 minutes each, totaling 12 sessions over 4 weeks).
  Interventions: Behavioral: Active Comparator #1

INTERVENTIONS:
Behavioral: Experimental Cognitive training in Immersive Virtual Reality and Telemedicine approach — The cognitive training involved a 4-week immersive virtual reality program to improve planning, cognitive flexibility, and information updating in patients with mild cognitive impairment related to Parkinson's disease. Over 12 sessions of 30 minutes each, participants trained in a virtual supermarket to strengthen attentional and executive skills. The planning task required creating and following a route to collect items while following rules, with increasing complexity. The cognitive flexibility task involved alternating between selecting items from different categories, with difficulty rising due to more categories and distractors. The updating task, set at a virtual checkout, challenged participants to memorize and recall items on a conveyor belt, with difficulty increasing based on sequence length and item count. Progression to higher levels required three successful trials, with feedback provided to support performance improvement
  Arms: Cognitive executive functions training implemented in immersive virtual reality, remotly delivered
Behavioral: Active Comparator #1 — The active placebo used the same virtual environment, Oculus Go system, and telemedicine setup as the training group, but engaged in tasks with low cognitive demands, mimicking everyday activities. The placebo-planning task involved following a fixed shopping list order in a modified version of the Zoo Map Test. The placebo-shifting task required selecting items from shelves without alternating between categories, while the placebo-updating task involved recalling only the last item from a conveyor belt sequence. The sessions mirrored the training group's structure, with 12 sessions over 4 weeks (3 per week, 30 minutes each), maintaining the same frequency, duration, and levels than Training.
  Arms: Active Placebo implemented in immersive virtual reality, remotly delivered

SUMMARY:
The goal of this randomized controlled trial is to evaluate the efficacy of attention and executive function training on prospective memory (PM) and executive functions in patients with Parkinson's disease and mild cognitive impairment (PD-MCI) and compare their performance to healthy volunteers. The study aims to determine whether immersive virtual reality (iVR) training can improve PM and executive function performance in PD-MCI patients, whether the effects of training are maintained over time, and how the PM and executive function performance of PD-MCI patients compares to that of healthy volunteers. Participants in the training group engage in real-life scenario exercises focused on planning, shifting, and updating tasks, while those in the placebo group perform simpler daily tasks with lower cognitive demands. Healthy volunteers serve as an additional control group. All sessions are conducted remotely using telemedicine and iVR headsets over a 4-week period. Outcome measures, including PM and executive function performance, are assessed at baseline, post-training, and a 2-month follow-up to evaluate the intervention's effectiveness and compare results across groups.

DETAILED DESCRIPTION:
This study examines the efficacy of attention and executive function training on prospective memory (PM) and executive functions in individuals with Parkinson's disease and mild cognitive impairment (PD-MCI), using a combined immersive virtual reality (iVR) and telemedicine approach. PM impairments, closely linked to deficits in episodic memory and executive functions, are a significant challenge in PD-MCI. Healthy volunteers are included as an additional group, undergoing the same intervention protocol, to evaluate baseline differences and the generalizability of the training effects.

Participants are randomly assigned to one of two arms: a training group (TR-C) or an active placebo group (AP-C). Both PD-MCI patients and healthy volunteers in the TR-C group engage in immersive virtual environments featuring real-life scenarios that require planning, task-switching, and updating skills, with tasks progressively increasing in complexity. The AP-C group completes simpler daily tasks with lower cognitive demands, serving as an active control condition. The intervention is conducted entirely remotely using telemedicine platforms and iVR headsets, ensuring accessibility and ecological validity. Assessments of PM and attention/executive functions are conducted at three time points: baseline (T0), post-training (T1, 4 weeks), and follow-up (T2, 2 months). The primary outcomes include improvements in PM performance and executive functions, as well as the retention of these training effects over time. By including healthy volunteers undergoing identical protocols, the study provides a robust comparison to evaluate both intervention-specific benefits and baseline cognitive differences between groups. This research aims to demonstrate the potential of iVR-based cognitive training to improve not only PM but also broader executive functions in both clinical and healthy populations, highlighting the applicability of innovative technologies in addressing cognitive challenges associated with neurodegenerative conditions and promoting cognitive health more broadly.

ELIGIBILITY:
Inclusion Criteria:

* PD-MCI: i) idiopathic PD, according with the United Kingdom Parkinson's disease Society brain bank criteria; ii) diagnosis of MCI from neuropsychological screening battery and MMSE; specifically, were included in the study PD-MCI whose performance was 1.5 standard deviations below the normative sample at least on two tests, one of which assessed executive functions; iii) absence of pronounced dyskinesia; iv) absence of other psychiatric and neurological disorders than PD; v) absence of other serious non-neurological disorders; vi) no treatment with deep brain stimulation. All patients had been stably treated with L-dopa and/or dopamine agonists for at least three months prior to the administration of the neuropsychological screening and outcome measures and throughout the duration of the entire experimental protocol.
* Healthy Volunteers: i) no neurologic or psychiatric illness; ii) no other disese than neurological; iii) no alchool abuse; iv) neuropsychological screening with rates between 3-4 equivalent score based on normative population

Exclusion Criteria:

* PD-MCI: i) Cognitive decline inconsistent with mild cognitive impairment; ii) no idiopathic Parkinson's disease; iii) presence of of important non neurological disease;
* Healthy volunteers: i) neuropsychological assessment characterized by a cognitive domain with a deficit or a score equivalent to 1 or 2, based on normative data; ii) presence of psychiatric or neurological disease

Ages: 56 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Prospective Memory Test | From baseline to Post-Training (4 weeks)
  Prospective memory was assessed using the Memory for Intentions Screening Test, a task designed to evaluate prospective memory through eight trials: four time-based and four event-based. Each trial reflects real-life scenarios, and participants perform an ongoing word search task simultaneously. Scores for prospective memory range from 0 (failure) to 2 (correct execution). The test includes a multiple-choice recognition task, scored from 0 to 1, with a total score ranging from 0 to 8. A 24-hour delayed task assesses the ability to recall and execute a planned action after a day, such as calling the examiner at a specific time and reporting sleep hours, with scores from 0 (failure) to 2 (successful execution).
Planning Tasks | From Baseline to Post-Training (4 weeks)
  All patients were administered neuropsychological tests at T0, T1 and T2.The assessment of planning skills were tested using the Zoo Map Test and Tower of London
Shifting Task | From Baseline to Post-Training (4 weeks)
  The assessment of shifting abilities were tested using the Trail Making Test and the Alternate Fluency Task
Updating task | From the baseline to Post-Training (4 weeks)
  All patients were administered neuropsychological tests at T0, T1 and T2.The assessment of updating was tested using the updating task belonging to the Zimmermann's Test of Every Day Attention.

SECONDARY OUTCOMES:
Effects duration over time | From the end of the training to 2-month follow-up
  Prospective Memory test (MIST) at 2-months follow up, (T2)

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Lucia Foundation, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available